CLINICAL TRIAL: NCT00026312
Title: Phase III Randomized Study of Chimeric Antibody 14.18 (Ch14.18) in High Risk Neuroblastoma Following Myeloablative Therapy and Autologous Stem Cell Rescue
Brief Title: Isotretinoin With or Without Dinutuximab, Aldesleukin, and Sargramostim Following Stem Cell Transplant in Treating Patients With Neuroblastoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01064; NCI-2009-01064 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s14-01661; COG-ANBL0032; PANBL0032_A33PAMDREVW01; CDR0000069018; ANBL0032; ANBL0032 (Other: Children's Oncology Group); ANBL0032 (Other: CTEP); U10CA030969 (NIH); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-06

CONDITIONS: Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Recurrent Neuroblastoma; Regional Neuroblastoma; Stage 4 Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — aldesleukin; dinutuximab; Isotretinoin; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (isotretinoin) (closed to accrual as of 4/16/2009) (Active Comparator): Beginning preferably between day 56 and day 85 post-ASCT, but may be delayed up to day 200, patients receive isotretinoin PO BID for 14 days. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients may cross over to Arm II provided they have not experienced disease progression and have not received any further anti-neuroblastoma therapy following completion of isotretinoin therapy.
  Interventions: Drug: Isotretinoin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment
- Arm II (sargramostim, dinutuximab, aldesleukin, isotretinoin) (Experimental): Beginning preferably between day 56 and day 85 post-ASCT, but may be delayed up to day 200, patients receive immunotherapy comprising sargramostim SC or IV over 2 hours on days 0-13 during courses 1, 3, and 5 and dinutuximab IV over 10-20 hours on days 3-6 of courses 1-5. Patients also receive aldesleukin IV continuously on days 0-3 and 7-10 during courses 2 and 4. Immunotherapy repeats every 28 days for 5 courses in the absence of disease progression or unacceptable toxicity. Patients also receive isotretinoin as in Arm I beginning on day 11 of immunotherapy.
  Interventions: Biological: Aldesleukin; Biological: Dinutuximab; Drug: Isotretinoin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Biological: Sargramostim

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
  Arms: Arm II (sargramostim, dinutuximab, aldesleukin, isotretinoin)
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; Dinutuximab Beta; MOAB Ch14.18; monoclonal antibody Ch14.18; Qarziba; Unituxin
  Arms: Arm II (sargramostim, dinutuximab, aldesleukin, isotretinoin)
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Absorica; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Myorisan; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret; ZENATANE
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Sargramostim — Given IV or SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
  Arms: Arm II (sargramostim, dinutuximab, aldesleukin, isotretinoin)

SUMMARY:
This partially randomized phase III trial studies isotretinoin with dinutuximab, aldesleukin, and sargramostim to see how well it works compared to isotretinoin alone following stem cell transplant in treating patients with neuroblastoma. Drugs used in chemotherapy, such as isotretinoin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as dinutuximab, may block tumor growth in different ways by targeting certain cells. Aldesleukin and sargramostim may stimulate a person's white blood cells to kill cancer cells. It is not yet known if chemotherapy is more effective with or without dinutuximab, aldesleukin, and sargramostim following stem cell transplant in treating neuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if monoclonal antibody Ch14.18 (dinutuximab) + cytokines + isotretinoin (13-cis-retinoic acid, or RA) improves event free survival after myeloablative therapy and stem cell rescue as compared to RA alone, in high risk neuroblastoma patients who have achieved a pre-autologous stem cell transplant (ASCT) response of complete response (CR), very good partial response (VGPR), or partial response (PR).

SECONDARY OBJECTIVES:

I. Determine if monoclonal antibody Ch14.18 + cytokines + isotretinoin (13-cis-retinoic acid, or RA) improves overall survival after myeloablative therapy and stem cell rescue as compared to RA alone, in high risk neuroblastoma patients who have achieved a pre-ASCT response of CR, VGPR, or PR.

II. Determine if immunotherapy + RA improves event free survival and overall survival as compared to RA alone, in the subgroup of high risk International Neuroblastoma Staging System (INSS) stage 4 neuroblastoma patients who have achieved a pre-ASCT response of CR, VGPR, or PR.

III. Determine the toxicities of the combination of monoclonal antibody Ch14.18 with cytokines.

IV. To compare the outcome data of the patients with persistent disease documented by biopsy (Stratum 07) to the historical data for the analogous patients from Children's Cancer Group (CCG)-3981.

V. To further describe and refine the event free survival (EFS) and overall survival (OS) estimates and baseline characteristics for subjects receiving Ch14.18 + cytokines + RA, following cessation of the randomized portion of the study.

VI. To further describe the safety and toxicity of Ch14.18 + cytokines + RA under the new administration guidelines implemented following cessation of the randomized portion of the study with focus on: a) number of courses delivered per subject; b) number of dose reductions or stoppage (ch14.18 and/or interleukin [IL]-2); and c) number of toxic deaths.

TERTIARY OBJECTIVES:

I. In the subgroup of neuroblastoma patients who have achieved a pre-ASCT response of CR, VGPR, or PR, determine if there is a difference between the two randomized regimens in reducing the minimal residual disease (MRD) burden as detected by the following parameters: meta-iodobenylguanidine (MIBG) scan, immunocytology (IC) of blood and bone marrow samples, reverse transcriptase-polymerase chain reaction (RT-PCR) for tyrosine hydroxylase, phosphoglycolate phosphatase (PGP) 9.5, and melanoma antigen family A, 1 (MAGE-1) in blood and bone marrow.

II. Determine if change from baseline of MRD is associated with event free and overall survival.

III. Determine whether tumor biology at diagnosis correlates with event-free and overall survival, for either of the randomized regimens.

IV. To explore the relationship between antibody-dependent cellular cytoxicity (ADCC) and EFS.

V. To determine a descriptive profile of human anti-chimeric antibody (HACA) during immunotherapy.

VI. To determine the variability of 13-cis-retinoic-acid pharmacokinetics and relationship to pharmacogenomic parameters and determine if these levels and/or genetic variations correlate with EFS or systemic toxicity.

VII. To determine the potential effect of ch14.18 on cardiac repolarization and to evaluate ch14.18 plasma levels.

VIII. To determine if the presence of naturally occurring anti-glycan antibodies correlates with allergic reactions and blood levels of ch14.18.

IX. To determine if the genotype of Fc receptor (FcR) and killer cell immunoglobulin-like receptor (Kir)/Kir-ligand correlate with EFS.

X. To determine if natural killer cell p30-related protein (NKp30) isoform expression and single nucleotide polymorphism (SNP), and circulating ligand B7-H6 are prognostic of EFS or OS.

OUTLINE: Patients stratified with biopsy-confirmed post-ASCT persistent disease who are also enrolled on Children's Oncology Group (COG)-A3973 or COG-ANBL0532 are assigned to treatment Arm II. Patients in the first set of strata are randomized to 1 of 2 treatment arms.

ARM I: Beginning on day 56-85 post-ASCT, patients receive isotretinoin orally (PO) twice daily (BID) for 14 days. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients may cross over to Arm II provided they have not experienced disease progression and have not received any further anti-neuroblastoma therapy following completion of isotretinoin therapy. (closed to accrual as of 4/16/2009)

ARM II: Beginning on day 56-85 post-ASCT, patients receive immunotherapy comprising sargramostim (GM-CSF) subcutaneously (SC) or intravenously (IV) over 2 hours on days 0-13 during courses 1, 3, and 5 and dinutuximab IV over 10-20 hours on days 3-6 of courses 1-5. Patients also receive aldesleukin IV continuously on days 0-3 and 7-10 during courses 2 and 4. Immunotherapy repeats every 28 days for 5 courses in the absence of disease progression or unacceptable toxicity. Patients also receive isotretinoin as in Arm I beginning on day 11 of immunotherapy.

After completion of study treatment, patients are followed up periodically for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be diagnosed with neuroblastoma, and categorized as high risk at the time of diagnosis; exception: patients who are initially diagnosed as non-high-risk neuroblastoma, but later converted (and/or relapsed) to high risk neuroblastoma are also eligible
* All patients must have completed therapy including intensive induction followed by ASCT and radiotherapy to be eligible for ANBL0032; radiotherapy may be waived for patients who either have small adrenal masses which are completely resected up front, or who never have an identifiable primary tumor; examples of such therapies include:

  * Following treatment per A3973 protocol
  * Following treatment per Pediatric Oncology Group (POG)-9341/9342 protocol
  * Following treatment per CCG3891
  * Following treatment on New Approaches to Neuroblastoma Therapy (NANT) 2001-02
  * Enrollment on or following treatment per ANBL02P1
  * Enrollment on or following treatment per ANBL07P1
  * Tandem transplant patients are eligible:

    * Following treatment on or per ANBL0532
    * Following treatment per POG 9640
    * Following treatment per COG ANBL00P1
    * Following treatment per CHP 594/Dana-Farber Cancer Institute (DFCI) 34-DAT
* No more than 12 months from the date of starting the first induction chemotherapy after diagnosis to the date of ASCT except for the rare occasions as noted below; for tandem ASCT patients, this will be the date of the FIRST stem cell infusion; exception: for those who are initially diagnosed as non-high risk neuroblastoma, but later converted (and/or relapsed) to high risk neuroblastoma, the 12 months restriction should start from the date of induction therapy for high risk neuroblastoma (not from the initial induction therapy for non-high risk disease), to the date of ASCT
* At pre-ASCT evaluation patients must meet the International Neuroblastoma Response Criteria (INRC) for CR, VGPR, or PR for primary site, soft tissue metastases and bone metastases; patients who meet those criteria must also meet the protocol specified criteria for bone marrow response as outlined below:

  * =< 10% tumor (of total nucleated cellular content) seen on any specimen from a bilateral bone marrow aspirate/biopsy
  * Patient who have no tumor seen on the prior bone marrow, and then have =< 10% tumor on any of the bilateral marrow aspirate/biopsy specimens done at pre-ASCT and/or pre-enrollment evaluation will also be eligible (note that per INRC this would have been defined as "overall" response of progressive disease [PD])
* Prior to enrollment on ANBL0032, a determination of mandatory disease staging must be performed (tumor imaging studies including computed tomography [CT] or magnetic resonance imaging [MRI], MIBG scan, and vanillylmandelic acid [VMA]/homovanillic acid [HVA]; bone marrow aspirates are required but biopsy may be omitted if negative prior to ASCT); this disease assessment is required for eligibility and should be done preferably within 2 weeks, but must be done within a maximum of 4 weeks before enrollment

  * For those with residual disease before radiotherapy, re-evaluation of irradiated residual tumors is preferably performed at the earliest 5 days after completing radiotherapy; patients with residual disease are eligible; biopsy is not required; patients who have biopsy proven residual disease after ASCT will be enrolled on Stratum 07
  * Patients must not have progressive disease at the time of study enrollment except for protocol specified bone marrow response and except for elevations of catecholamines as the only sign of disease in a patient who had normal catecholamines at pre-ASCT evaluation
* Patients must be enrolled before treatment begins; the date protocol therapy is projected to start must be no later than ten (10) calendar days after the date of study enrollment; patients should be enrolled preferably between day 56 and day 85 after peripheral blood stem cell (PBSC) infusion (day from 2nd stem cell infusion for tandem transplant); patients must be enrolled no later than day 200 after PBSC infusion; enrollment must occur after completion of radiotherapy, and after completion of tumor assessment post-ASCT and radiotherapy; informed consent should be obtained within 3 weeks pre-ASCT up to the time of registration
* Patients must not have received prior anti-disialoganglioside (GD2) antibody therapy
* Patients must have a Lansky or Karnofsky performance scale score of >= 50% and patients must have a life expectancy of >= 2 months
* Total absolute phagocyte count (APC = %neutrophils + %monocytes) X white blood cell (WBC) is at least 1000/uL
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * No greater than 0.4 mg/dL (1 month to < 6 months)
  * No greater than 0.5 mg/dL (6 months to < 1 year)
  * No greater than 0.6 mg/dL (1 to < 2 years)
  * No greater than 0.8 mg/dL (2 to < 6 years)
  * No greater than 1.0 mg/dL (6 to < 10 years)
  * No greater than 1.2 mg/dL (10 to < 13 years)
  * No greater than 1.4 mg/dL (>= 13 years [female])
  * No greater than 1.5 mg/dL (13 to < 16 years [male])
  * No greater than 1.7 mg/dL (>= 16 years [male])
* Total bilirubin =< 1.5 x normal
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 5 x normal
* Veno-occlusive disease, if present, should be stable or improving
* Shortening fraction of >= 27% by echocardiogram, or if shortening fraction abnormal, ejection fraction of >= 55% by gated radionuclide study or echocardiogram; note: the echocardiogram or gated radionuclide study must be performed within 4 weeks prior to enrollment
* Forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) > 60% predicted by pulmonary function test; for children who are unable to do pulmonary function tests (PFTs), no evidence of dyspnea at rest and no exercise intolerance should be documented; note: the pulmonary function test must be performed within 4 weeks prior to enrollment
* Patients with seizure disorder may be enrolled if on anticonvulsants and well-controlled; central nervous system (CNS) toxicity < grade 2
* Written informed consent in accordance with institutional and Food and Drug Administration (FDA) guidelines must be obtained from parent or legal guardian
* Females of childbearing potential must have a negative pregnancy test; patients of childbearing potential must agree to use an effective birth control method; female patients who are lactating must agree to stop breast-feeding

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1449 (Actual)
Dates: Start 2001-10-18 (Actual); Primary Completion 2012-01-12 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alice L Yu, Principal Investigator — Children's Oncology Group
Locations (197):
- United States (172):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Oesterheld J, Ferguson W, Kraveka JM, Bergendahl G, Clinch T, Lorenzi E, Berry D, Wada RK, Isakoff MS, Eslin DE, Brown VI, Roberts W, Zage P, Harrod VL, Mitchell DS, Hanson D, Saulnier Sholler GL. Eflornithine as Postimmunotherapy Maintenance in High-Risk Neuroblastoma: Externally Controlled, Propensity Score-Matched Survival Outcome Comparisons. J Clin Oncol. 2024 Jan 1;42(1):90-102. doi: 10.1200/JCO.22.02875. Epub 2023 Oct 26. PMID 37883734
- [Derived] Desai AV, Gilman AL, Ozkaynak MF, Naranjo A, London WB, Tenney SC, Diccianni M, Hank JA, Parisi MT, Shulkin BL, Smith M, Moscow JA, Shimada H, Matthay KK, Cohn SL, Maris JM, Bagatell R, Sondel PM, Park JR, Yu AL. Outcomes Following GD2-Directed Postconsolidation Therapy for Neuroblastoma After Cessation of Random Assignment on ANBL0032: A Report From the Children's Oncology Group. J Clin Oncol. 2022 Dec 10;40(35):4107-4118. doi: 10.1200/JCO.21.02478. Epub 2022 Jul 15. PMID 35839426
- [Derived] Yu AL, Gilman AL, Ozkaynak MF, London WB, Kreissman SG, Chen HX, Smith M, Anderson B, Villablanca JG, Matthay KK, Shimada H, Grupp SA, Seeger R, Reynolds CP, Buxton A, Reisfeld RA, Gillies SD, Cohn SL, Maris JM, Sondel PM; Children's Oncology Group. Anti-GD2 antibody with GM-CSF, interleukin-2, and isotretinoin for neuroblastoma. N Engl J Med. 2010 Sep 30;363(14):1324-34. doi: 10.1056/NEJMoa0911123. PMID 20879881

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A: Randomized to Regimen A - RA Only
- Regimen B: Regimen B - RA + Immunotherapy
Period: Overall Study
Arm/Group | Regimen A | Regimen B
Started | 116 | 1333
Completed | 82 | 1064
Not Completed | 34 | 269
Not completed — Adverse Event | 0 | 32
Not completed — Death | 1 | 7
Not completed — Lack of Efficacy | 19 | 114
Not completed — Lost to Follow-up | 0 | 5
Not completed — Physician Decision | 1 | 37
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Ineligible | 4 | 5
Not completed — Entry onto another COG study | 0 | 1
Not completed — Refusal by patient/parent/guardian | 8 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A | Regimen B | Total
Number analyzed (Participants) | 116 | 1333 | 1449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 116 | 1325 | 1441
  Between 18 and 65 years | 0 | 8 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.22 (2.12) | 3.64 (2.77) | 3.61 (2.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 534 | 583
  Male | 67 | 799 | 866
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 142 | 153
  Not Hispanic or Latino | 99 | 1159 | 1258
  Unknown or Not Reported | 6 | 32 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 4 | 62 | 66
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 8 | 153 | 161
  White | 89 | 942 | 1031
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 171 | 184
Region of Enrollment [Number; unit: participants]
  New Zealand | 0 | 17 | 17
  Canada | 13 | 135 | 148
  United States | 100 | 1092 | 1192
  Australia | 3 | 89 | 92

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS)
Description: Comparison to determine if RA + Immunotherapy improves EFS as compared to RA Only
Time Frame: Three years
Population: Eligible, randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Regimen B: Randomized to Regimen B - RA + Immunotherapy
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 112 | 114
Percentage of participants | 48.1 [38.4 to 57.8] | 62.9 [54.0 to 71.9]
Statistical Analysis 1: Comparison: Regimen A vs Regimen B; The event-free survival distributions of patients randomized to Regimen A - RA Only and randomized to Regimen B - RA + Immunotherapy were compared using the log-rank test; Test type: Superiority or Other; p = 0.1016, Log Rank; Log Rank Test Statistic = 2.6803

2. Secondary Outcome: Event-Free Survival (EFS)
Description: Comparison to determine if RA + Immunotherapy improves EFS as compared to RA Only for the subgroup of randomized patients with INSS Stage 4 disease. Descriptive comparison of outcome data for patients with persistent disease documented by biopsy to historical data for the analogous patients from CCG-3981.
Time Frame: Three years
Population: Eligible, randomized patients with INSS Stage 4 disease. Eligible patients with persistent disease.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 93 | 127
Percentage of participants
  Randomized patients with INSS Stage 4 disease: number analyzed (Participants) | 93 | 90
  Randomized patients with INSS Stage 4 disease | 43.2 [32.5 to 53.8] | 59.7 [49.5 to 69.9]
  Eligible patients with persistent disease: number analyzed (Participants) | 0 | 37
  Eligible patients with persistent disease |  | 35.1 [19.8 to 50.5]
Statistical Analysis 1: Comparison: Regimen A vs Regimen B; The event-free survival distributions of patients randomized to Regimen A - RA Only and randomized to Regimen B - RA + Immunotherapy for the subgroup of patients with INSS Stage 4 disease were compared using the log-rank test; Test type: Superiority or Other; p = 0.1057, Log Rank; Log Rank Test Statistic = 2.6176

3. Secondary Outcome: Event-Free Survival (EFS) of Patients From the Non-randomized Portion of the Trial
Description: EFS for patients receiving RA + Immunotherapy following the cessation of the randomized portion of the study.
Time Frame: Three years
Population: Eligible patients non-randomly assigned to Regimen B after halting of randomization, excluding patients with persistent disease.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Regimen B: Non-randomly assigned to Regimen B after halting of randomization, excluding patients with persistent disease
Arm/Group | Regimen B
Number analyzed (Participants) | 1177
Percentage of participants | 64.0 [60.2 to 67.8]

4. Secondary Outcome: Incidence of Toxicities Assessed Using Common Terminology Criteria for Adverse Events Version 4.0
Description: Proportion of patients experiencing at least one Grade 3 or higher toxicity.
Time Frame: From enrollment to follow-up
Population: Eligible patients enrolled prior to halting of randomization.
Measure: Number (95% Confidence Interval); unit: Proportion
Groups:
- Regimen B: Patients that received RA + Immunotherapy before halting of randomization
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 112 | 141
Proportion | 0.64 [0.55 to 0.73] | 0.94 [0.90 to 0.98]

5. Secondary Outcome: Number of Courses of Therapy Delivered
Description: Number of courses of therapy delivered for patients randomized to RA + Immunotherapy vs. patients non-randomly assigned to RA + Immunotherapy, excluding patients with persistent disease.
Time Frame: Courses 1-6
Population: Eligible patients assigned to Regimen B, excluding patients with persistent disease.
Measure: Median (Full Range); unit: courses per patient
Groups:
- Regimen B: Regimen B- RA + Immunotherapy
Arm/Group | Regimen B
Number analyzed (Participants) | 1291
courses per patient
  Randomized to Regimen B - RA + Immunotherapy | 6 [0 to 6]
  Non-randomly assigned after halting randomization | 6 [0 to 6]
Statistical Analysis 1: Comparison: Regimen B; The number of courses of therapy delivered or patients randomized to Regimen B - RA + Immunotherapy and non-randomly assigned to Regimen B after halting of randomization, excluding patients with persistent disease, were compared using the Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.0262, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0

6. Secondary Outcome: Overall Survival (OS)
Description: Comparison to determine if RA + Immunotherapy improves OS as compared to RA Only. Comparison to determine if RA + Immunotherapy improves OS as compared to RA only and for the subgroup of randomized patients with INSS Stage 4 disease.
Time Frame: Three years
Population: Eligible, randomized patients. Eligible, randomized patients with INSS Stage 4 disease.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 112 | 114
Percentage of participants
  Randomized patients | 67.4 [58.3 to 76.5] | 78.8 [71.2 to 86.4]
  Randomized patients with INSS Stage 4 disease: number analyzed (Participants) | 93 | 90
  Randomized patients with INSS Stage 4 disease | 64.0 [53.8 to 74.3] | 78.7 [70.2 to 87.2]
Statistical Analysis 1: Comparison: Regimen A vs Regimen B; The overall survival distributions of patients randomized to Regimen A - RA Only and randomized to Regimen B - RA + Immunotherapy were compared using the log-rank test; Test type: Superiority or Other; p = 0.0634, Log Rank; Log Rank Test Statistic = 3.4471
Statistical Analysis 2: Comparison: Regimen A vs Regimen B; The overall survival distributions of patients randomized to Regimen A - RA Only and randomized to Regimen B - RA + Immunotherapy for the subgroup of patients with INSS Stage 4 disease were compared using the log-rank test; Test type: Superiority or Other; p = 0.042, Log Rank; Log-Rank Test Statistic = 4.1362

7. Secondary Outcome: Overall Survival (OS) of Patients From the Non-randomized Portion of the Trial
Description: OS for patients receiving RA + Immunotherapy following the cessation of the randomized portion of the study.
Time Frame: Three years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen B
Number analyzed (Participants) | 1177
Percentage of participants | 78.4 [75.1 to 81.6]

8. Other Pre Specified Outcome: Average Level of HACA
Description: The average level of HACA at each collection time point during immunotherapy will be calculated.
Time Frame: Up to 10 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Cardiac Repolarization
Description: In general, descriptive summaries will include n, mean, standard deviation, median, minimum, maximum and 90% confidence intervals for continuous variables, and n and percent for categorical variables. Summaries will present data by assessment time when appropriate.
Time Frame: Up to 10 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in MRD
Description: A descriptive analysis of the change from baseline of MRD will be performed. Also, a Wilcoxon rank-sum test will be performed to compare the median change from baseline of MRD between the two treatment arms. A multivariate Cox proportional hazards regression model will test to see if the change in MRD burden is associated with EFS or OS.
Time Frame: Baseline to up to 10 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Tumor Biology
Description: A multivariate Cox proportional hazards regression model will test to see if the dinutuximab serum level, HACA titer, effector cell function, or serum marker for effector cell activation are associated with EFS or OS.
Time Frame: Baseline to up to 10 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Circulating B7-H6 Levels
Description: Kaplan-Meier plots of EFS and OS will be generated after dichotomization using the median value for the cohort. To determine the prognostic value of circulating B7-H6 level, univariate analysis will be performed using a log rank test for EFS and OS. In multivariable analysis of EFS and OS, Cox models will be used to test for the independent prognostic ability of circulating B7-H6 level, adjusting for significant prognostic factors including MYCN status, INSS stage, histology and age at diagnosis.
Time Frame: 1 week before first sargramostim injection (day -1 of course 1)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Genotype of FcR
Description: Kaplan-Meier plots of EFS will be generated for the three genotype subgroups of FcR as well as for the three genotype subgroups of Kir/Kir-ligand. In addition, a log rank test comparison will be made in a pairwise fashion of each of the genotypes within FcR and within Kir/Kir-ligand.
Time Frame: Up to 10 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Genotype of Kir/Kir-ligand
Description: as for outcome 13
Time Frame: Up to 10 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Isotretinoin Pharmacokinetic Parameters
Description: To determine if there is a relationship of the peak serum concentration level with EFS, the term for this level will be tested in a Cox proportional hazards model. To determine if there is a relationship of the peak serum concentration level with toxicity rates, Kendall's Tau statistic will be calculated.
Time Frame: At 4 hours after administration on day 14 of course 1
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Levels of ADCC
Description: Will be descriptively compared.
Time Frame: Up to 10 years
Reporting Status: Not Posted

17. Other Pre Specified Outcome: NKp30 Isoform Expression and SNP
Description: Kaplan-Meier plots of EFS and OS will be generated after dichotomization using the median value for the cohort. To determine the prognostic value of NKp30 isoform expression and SNP, univariate analysis will be performed using a log rank test for EFS and OS. In multivariable analysis of EFS and OS, Cox models will be used to test for the independent prognostic ability of NKp30 isoform expression and SNP, adjusting for significant prognostic factors including v-MYC myelocytomatosis viral related oncogene, neuroblastoma derived (avian) (MYCN) status, INSS stage, histology and age at diagnosis.
Time Frame: 1 week before first sargramostim injection (day -1 of course 1)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Presence of Naturally Occurring Anti-glycan Antibodies
Description: A Fisher's exact test will be performed to determine if the presence of naturally occurring anti-glycan antibodies correlates with allergic reactions. A Wilcoxon test will be performed to determine if the presence of naturally occurring anti-glycan antibodies correlates with blood levels of dinutuximab.
Time Frame: Up to 10 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Ineligible patients were excluded from the adverse event analysis, so only eligible patients are reported.
Arm/Group | Regimen A | Regimen B
Serious Adverse Events (participants affected / at risk) | 10/112 | 785/1328
Other Adverse Events (participants affected / at risk) | 92/112 | 1244/1328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (N=112) | Regimen B (N=1328)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 42 (49)
Blood and lymphatic system disorders - Other specify (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac disorders - Other specify (Cardiac disorders) | 1 (1) | 5 (5)
Heart failure (Cardiac disorders) | 0 (0) | 3 (3)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 7 (7)
Pericardial effusion (Cardiac disorders) | 0 (0) | 3 (3)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 13 (16)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Ear and labyrinth disorders - Other specify (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Endocrine disorders - Other specify (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 4 (4)
Blurred vision (Eye disorders) | 0 (0) | 7 (7)
Eye disorders - Other specify (Eye disorders) | 1 (1) | 16 (16)
Optic nerve disorder (Eye disorders) | 0 (0) | 2 (2)
Papilledema (Eye disorders) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 0 (0) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 41 (60)
Ascites (Gastrointestinal disorders) | 0 (0) | 5 (5)
Colitis (Gastrointestinal disorders) | 0 (0) | 9 (10)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 35 (36)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 10 (10)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 4 (4)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 14 (16)
Chills (General disorders) | 0 (0) | 5 (5)
Death NOS (General disorders) | 0 (0) | 3 (3)
Edema face (General disorders) | 0 (0) | 12 (13)
Edema limbs (General disorders) | 0 (0) | 2 (2)
Edema trunk (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 8 (8)
Fever (General disorders) | 0 (0) | 121 (148)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other specify (General disorders) | 0 (0) | 4 (4)
Infusion related reaction (General disorders) | 0 (0) | 4 (4)
Injection site reaction (General disorders) | 0 (0) | 2 (2)
Irritability (General disorders) | 0 (0) | 6 (6)
Localized edema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 6 (6)
Pain (General disorders) | 0 (0) | 47 (68)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (3) | 141 (185)
Anaphylaxis (Immune system disorders) | 1 (1) | 153 (180)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 23 (35)
Immune system disorders - Other specify (Immune system disorders) | 0 (0) | 1 (1)
Serum sickness (Immune system disorders) | 0 (0) | 5 (7)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Bone infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 88 (105)
Device related infection (Infections and infestations) | 0 (0) | 4 (4)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 11 (11)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other specify (Infections and infestations) | 0 (0) | 113 (145)
Kidney infection (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 13 (14)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 33 (35)
Skin infection (Infections and infestations) | 0 (0) | 4 (4)
Upper respiratory infection (Infections and infestations) | 0 (0) | 9 (10)
Urinary tract infection (Infections and infestations) | 0 (0) | 11 (13)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (3) | 36 (45)
Alkaline phosphatase increased (Investigations) | 0 (0) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 28 (30)
Blood bilirubin increased (Investigations) | 0 (0) | 21 (21)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 14 (15)
Fibrinogen decreased (Investigations) | 0 (0) | 2 (2)
GGT increased (Investigations) | 0 (0) | 14 (18)
INR increased (Investigations) | 0 (0) | 2 (2)
Investigations - Other specify (Investigations) | 0 (0) | 5 (5)
Lipase increased (Investigations) | 0 (0) | 3 (3)
Lymphocyte count decreased (Investigations) | 2 (2) | 17 (22)
Neutrophil count decreased (Investigations) | 0 (0) | 30 (31)
Platelet count decreased (Investigations) | 0 (0) | 29 (44)
Serum amylase increased (Investigations) | 0 (0) | 2 (2)
Urine output decreased (Investigations) | 0 (0) | 27 (37)
Weight gain (Investigations) | 0 (0) | 8 (8)
Weight loss (Investigations) | 0 (0) | 5 (6)
White blood cell decreased (Investigations) | 0 (0) | 15 (17)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 10 (10)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 16 (18)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 22 (22)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 24 (35)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 10 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 23 (25)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 23 (25)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 65 (71)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 66 (76)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 38 (40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal and connective tissue disorder - Other specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 20 (29)
Neoplasms benign malignant and unspecified (incl cysts and polyps) - Other specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 7 (7)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 3 (3)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 11 (12)
Hydrocephalus (Nervous system disorders) | 0 (0) | 4 (4)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 6 (6)
Myelitis (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other specify (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 11 (12)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 5 (5)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 10 (10)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Euphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 12 (12)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 9 (12)
Renal and urinary disorders - Other specify (Renal and urinary disorders) | 0 (0) | 3 (4)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 10 (11)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 11 (12)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 30 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 16 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 53 (60)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 69 (85)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (8)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (10)
Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 10 (10)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Skin and subcutaneous tissue disorders - Other specify (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 102 (128)
Surgical and medical procedures - Other specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 154 (189)
Hypertension (Vascular disorders) | 0 (0) | 22 (24)
Hypotension (Vascular disorders) | 0 (0) | 249 (335)
Thromboembolic event (Vascular disorders) | 0 (0) | 4 (4)
Vascular disorders - Other specify (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (N=112) | Regimen B (N=1328)
Anemia (Blood and lymphatic system disorders) | 22 (47) | 428 (962)
Blood and lymphatic system disorders - Other specify (Blood and lymphatic system disorders) | 1 (1) | 16 (24)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 19 (23)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other specify (Cardiac disorders) | 1 (1) | 36 (49)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 2 (2)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mobitz type I (Cardiac disorders) | 0 (0) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 5 (6)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 49 (82)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 8 (13)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Ear and labyrinth disorders - Other specify (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 3 (3)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 6 (8) | 22 (28)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 3 (3)
Endocrine disorders - Other specify (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 4 (6)
Hypothyroidism (Endocrine disorders) | 2 (2) | 6 (6)
Blurred vision (Eye disorders) | 0 (0) | 12 (14)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 2 (2)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other specify (Eye disorders) | 2 (2) | 20 (24)
Eye pain (Eye disorders) | 0 (0) | 2 (3)
Flashing lights (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 2 (3) | 8 (8)
Watering eyes (Eye disorders) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 11 (14) | 312 (566)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Cheilitis (Gastrointestinal disorders) | 4 (7) | 16 (29)
Colitis (Gastrointestinal disorders) | 0 (0) | 11 (14)
Colonic stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 24 (35)
Diarrhea (Gastrointestinal disorders) | 16 (26) | 196 (311)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 0 (0) | 5 (6)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (6)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 3 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 2 (5)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 40 (65)
Oral pain (Gastrointestinal disorders) | 0 (0) | 8 (9)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 4 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 4 (4)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 16 (23)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 21 (35) | 109 (196)
Chills (General disorders) | 0 (0) | 31 (43)
Edema face (General disorders) | 0 (0) | 49 (82)
Edema limbs (General disorders) | 0 (0) | 20 (28)
Edema trunk (General disorders) | 0 (0) | 3 (3)
Facial pain (General disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 2 (3) | 33 (39)
Fever (General disorders) | 33 (43) | 536 (991)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 4 (4)
General disorders and administration site conditions - Other specify (General disorders) | 0 (0) | 6 (8)
Hypothermia (General disorders) | 0 (0) | 2 (2)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 10 (13)
Irritability (General disorders) | 0 (0) | 13 (17)
Localized edema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 10 (12)
Pain (General disorders) | 6 (14) | 441 (941)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 0 (0) | 3 (3)
Allergic reaction (Immune system disorders) | 11 (29) | 655 (1405)
Anaphylaxis (Immune system disorders) | 1 (2) | 71 (92)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 115 (205)
Immune system disorders - Other specify (Immune system disorders) | 0 (0) | 4 (4)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 2 (2) | 8 (11)
Anorectal infection (Infections and infestations) | 0 (0) | 4 (4)
Bladder infection (Infections and infestations) | 0 (0) | 2 (2)
Bone infection (Infections and infestations) | 0 (0) | 3 (3)
Bronchial infection (Infections and infestations) | 2 (2) | 1 (1)
Catheter related infection (Infections and infestations) | 8 (9) | 97 (128)
Cecal infection (Infections and infestations) | 0 (0) | 2 (2)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 7 (8)
Endocarditis infective (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 39 (47)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 1 (1) | 1 (1)
Infections and infestations - Other specify (Infections and infestations) | 29 (42) | 147 (255)
Joint infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 13 (13)
Lymph gland infection (Infections and infestations) | 1 (1) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 6 (6)
Ovarian infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 3 (4)
Salivary gland infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 6 (6)
Sinusitis (Infections and infestations) | 1 (1) | 4 (4)
Skin infection (Infections and infestations) | 1 (1) | 9 (9)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory infection (Infections and infestations) | 2 (2) | 21 (23)
Urinary tract infection (Infections and infestations) | 1 (1) | 27 (35)
Wound infection (Infections and infestations) | 0 (0) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Injury poisoning and procedural complications - Other specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 6 (6)
Alanine aminotransferase increased (Investigations) | 33 (79) | 281 (560)
Alkaline phosphatase increased (Investigations) | 7 (14) | 35 (53)
Aspartate aminotransferase increased (Investigations) | 6 (11) | 180 (279)
Blood bilirubin increased (Investigations) | 5 (7) | 28 (40)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 1 (1)
Cholesterol high (Investigations) | 1 (4) | 12 (30)
Creatinine increased (Investigations) | 6 (12) | 44 (67)
Fibrinogen decreased (Investigations) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 97 (217)
INR increased (Investigations) | 0 (0) | 2 (2)
Investigations - Other specify (Investigations) | 2 (4) | 18 (28)
Lipase increased (Investigations) | 0 (0) | 4 (4)
Lymphocyte count decreased (Investigations) | 40 (97) | 323 (739)
Lymphocyte count increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 18 (24) | 272 (470)
Pancreatic enzymes decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 47 (144) | 356 (876)
Serum amylase increased (Investigations) | 0 (0) | 5 (12)
Urine output decreased (Investigations) | 0 (0) | 31 (57)
Weight gain (Investigations) | 0 (0) | 50 (90)
Weight loss (Investigations) | 0 (0) | 15 (15)
White blood cell decreased (Investigations) | 16 (37) | 158 (297)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 25 (48)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 5 (12) | 100 (189)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 14 (14)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 8 (17) | 36 (44)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5) | 77 (129)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 46 (58)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 13 (13)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 12 (12)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 11 (17) | 77 (162)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4) | 156 (359)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 128 (229)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 29 (35)
Hypokalemia (Metabolism and nutrition disorders) | 6 (12) | 409 (664)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 40 (55)
Hyponatremia (Metabolism and nutrition disorders) | 13 (31) | 262 (466)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (7) | 114 (141)
Iron overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (7) | 14 (18)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 69 (97)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 14 (17)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 16 (19)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal and connective tissue disorder - Other specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 9 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 26 (36)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7) | 132 (207)
Pelvic soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 7 (7)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (3)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 56 (73)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other specify (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 53 (119)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 4 (5) | 12 (17)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (4) | 19 (27)
Seizure (Nervous system disorders) | 1 (1) | 9 (9)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 2 (3) | 15 (20)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 3 (4)
Euphoria (Psychiatric disorders) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 0 (0) | 2 (2)
Personality change (Psychiatric disorders) | 4 (5) | 3 (3)
Psychosis (Psychiatric disorders) | 0 (0) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (2)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 17 (22)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 3 (6) | 32 (42)
Renal and urinary disorders - Other specify (Renal and urinary disorders) | 1 (2) | 10 (13)
Renal hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 30 (47)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (4)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 4 (4)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 2 (4)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 10 (12)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 5 (7)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 29 (36)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 84 (115)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 111 (146)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 179 (275)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (16)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (10)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (10)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 16 (29) | 57 (98)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 6 (7) | 6 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 13 (15)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 60 (89)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (8) | 41 (48)
Skin and subcutaneous tissue disorders - Other specify (Skin and subcutaneous tissue disorders) | 2 (2) | 22 (35)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 6 (9) | 606 (1151)
Capillary leak syndrome (Vascular disorders) | 2 (2) | 533 (1089)
Flushing (Vascular disorders) | 0 (0) | 5 (5)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 7 (16) | 48 (67)
Hypotension (Vascular disorders) | 6 (9) | 797 (1824)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Vascular disorders - Other specify (Vascular disorders) | 3 (5) | 17 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less